CLINICAL TRIAL: NCT01045382
Title: Co-transplantation of Mesenchymal Stem Cells and HLA-mismatched Allogeneic Hematopoietic Cells After Nonmyeloablative Conditioning: a Phase II Randomized Double-blind Study
Brief Title: MSC and HSC Coinfusion in Mismatched Minitransplants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment too slow
Sponsor: University of Liege (Other)
Collaborators: AZ Sint-Jan AV (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Jules Bordet Institute (Other); Universiteit Antwerpen (Other); AZ-VUB (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Yves Beguin, Prof, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJB0909
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoblastic, Acute; Leukemia, Myelocytic, Chronic; Myeloproliferative Disorders; Myelodysplastic Syndromes; Multiple Myeloma; Leukemia, Lymphocytic, Chronic; Hodgkin's Disease; Lymphoma, Non-Hodgkin
Keywords: HSC transplantation; HLA-mismatched; Mesenchymal stem cells; GVHD; co-infusion
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders; Myelodysplastic Syndromes; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Isotonic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mensenchymal Stem Cells (Experimental): Efficacy of MSC infusion on one-year overall survival of patients transplanted with HLA-mismatched PBSC.
  Patients will receive a conditioning regimen consisting in fludarabine (total dose 90 mg/square meter) and 2 Gy total body irradiation.
  MSC cells (1,5-3,0 x 10E6 MSC/Kg BW) will be injected, followed, at least one hour later, by the infusion of HLA-mismatched PBSC from related or unrelated donor.
  Interventions: Biological: Mesenchymal stem cells
- Placebo (Placebo Comparator): Patients will receive a conditioning regimen consisting in fludarabine (total dose 90 mg/square meter) and 2Gy total body irradiation.
  Isotonic solution will be injected will be injected, followed, at least one hour later, by the infusion of HLA-mismatched PBSC from related or unrelated donor.
  Interventions: Other: Isotonic solution

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal stem cell injection
  Arms: Mensenchymal Stem Cells
Other: Isotonic solution — Isotonic solution injection
  Arms: Placebo

SUMMARY:
The present project aims at evaluating the capacity of MSC to improve one-year overall survival of patients transplanted with HLA-mismatched PBSC from related or unrelated donors after non-myeloablative conditioning.

Co-infusion of MSC has been shown to facilitate engraftment of hematopoietic stem cell (HSC) in an immunodeficient mouse model. In addition, it has been shown that infusion of third party MSC in HSC transplantation could be successfully used as treatment for grade II-IV steroid-refractory acute graft versus host disease.

One hundred and twenty patients with HLA-mismatched donors will be included over 6 years at multiple centers across Belgium through the transplant committee of the Belgian Hematological Society. The conditioning regimen will consist of fludarabine and 2 Gy TBI, followed by the infusion of donor HSC. Patients will be randomized 1/1 in double-blind fashion to receive or not MSC (1.5-.3.0 x106/kg) from third-party (either haploidentical family members or unrelated volunteer) donors on day 0. Postgrafting immunosuppression will combine tacrolimus and MMF. Except for the collection, expansion and infusion of MSC, the clinical management of the patient will not differ from that of routine NM-HCT.

ELIGIBILITY:
Inclusion Criteria:

* Theoretical indication for a standard allo-transplant, but not feasible because: Age > 55 yrs. Unacceptable end organ performance. Patient's refusal.
* Indication for a standard auto-transplant: perform mini-allotransplantation 2-6 months after standard autotransplant.
* Male or female; fertile female patients must use a reliable contraception method
* Age ≤ 75 year old
* Informed consent given by patient or his/her guardian if of minor age.
* One or two HLA mismatches with PBSC:

  * One antigenic mismatch at HLA-A or -B or -C or -DRB1 or -DQB1
  * Two allelic mismatches at HLA-A or -B or -C or -DRB1 or -DQB1
  * One antigenic mismatch: 1 allelic mismatch at HLA-A or -B or -C or -DRB1 or -DQB1.
  * One antigenic mismatch at -DQB1 and one other antigenic mismatch at HLA-A or -B or -C or -DRB1
  * Patients with one single allelic mismatch at HLA-A or -B or -C or -DRB1 or -DQB1 can also be included in the protocol.
* Hematological malignancies confirmed histologically and not rapidly progressing:

  * AML in complete remission
  * ALL in complete remission
  * CML unresponsive/intolerant to Imatinib but not in blast crisis
  * Other myeloproliferative disorders not in blast crisis and not with extensive myelofibrosis
  * MDS with <5% blasts
  * Multiple myeloma not rapidly progressing
  * CLL
  * Non-Hodgkin's lymphoma (aggressive NHL should be chemosensitive)
  * Hodgkin's disease

Exclusion Criteria:

* Any condition not fulfilling inclusion criteria
* HIV positive
* Terminal organ failure, except for renal failure (dialysis acceptable)

  * Cardiac: Symptomatic coronary artery disease or other cardiac failure requiring therapy; ejection fraction <35%; uncontrolled arrhythmia; uncontrolled hypertension
  * Pulmonary: DLCO < 35% and/or receiving supplementary continuous oxygen
  * Hepatic: Fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease
* Uncontrolled infection, arrhythmia or hypertension
* Previous radiation therapy precluding the use of 2 Gy TBI
* 10/10 HLA-A, -B, -C, DRB1 and DQBI allele-matched donor fit to/willing to donate PBSC.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
One-year overall survival in the 2 arms. | One year

SECONDARY OUTCOMES:
Incidence of grade II-IV and grade III-IV acute GVDH | 100 days
Number of absolute donor T cells after HCT in each arm | 28
Cumulative incidence of non-relapse mortality | 100, 365 and 730 days
Incidence of extensive chronic GVHD in each arm | 365 days
Incidence of graft rejection in each arm. | 365 days
Quality and timing of immunologic reconstitution in each arm. | 100, 365 and 730 days
Detection of MSC from donor origin in recipient marrow after HCT in patients given MSC | 40 days
Proportion of patients with measurable disease at HCT who achieve a complete response in each arm. | 100, 365 and 730 days
Cumulative incidence of relapse | 365 and 730 days
Incidence of progression-free survival | 365 and 730 days
Incidence of infections | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Yves Beguin, MD, PhD, Principal Investigator — CHU-ULg; Frédéric Baron, MD, PhD, Study Chair — CHU-ULg; Evelyne Willems, MD, Principal Investigator — CHU-ULg; Dominik Selleslag, MD, PhD, Principal Investigator — AZ Brugge; Pierre Zachée, MD, PhD, Principal Investigator — ZNA Antwerpen; Philippe Lewalle, MD, PhD, Principal Investigator — Bordet Institute, Brussels; Dominique Bron, MD, PhD, Principal Investigator — Bordet Institute, Brussels; Wilfried Schroyens, MD, PhD, Principal Investigator — UZA Antwerpen; Chantal Lechanteur, PhD, Principal Investigator — CHU-ULg; Etienne Baudoux, MD, Principal Investigator — CHU-ULg; Johan Maertens, MD, Principal Investigator — KUL, Leuven; Rik Schots, MD, PhD, Principal Investigator — AZ VUB, Brussels; Augustin Ferrant, MD, PhD, Principal Investigator — UCL St. LUC, Brussels; Lucien Noens, MD, PhD, Principal Investigator — UZG Gent; Chantal Doyen, MD, PhD, Principal Investigator — Cliiques Universitaire Mont-Godinne, Yvoir; Tessa Kerre, MD, PhD, Principal Investigator — UZA, Antwerpen; Carlos Graux, MD, PhD, Principal Investigator — Cliniques Universitaires, Mont-Godinne
Locations (10):
- Belgium (10):
  - UZA, Edegem, Antwerpen
  - St-Luc UCL, Brussels, Brabant
  - AZ Gasthuisberg Leuven, Leuven, Flamish Brabant
  - UZ Gent, Ghent, Flanders Ost
  - AZ St-Jan, Bruges, Flanders West
  - Cliniques Universitaires Mont-Godinne, Yvoir, Namur
  - Hôpital Stuyvenberg, Antwerp
  - Bordet Institute, Brussels
  - Vrije Universiteit Brussel, Brussels
  - CHU-ULg, Liège